CLINICAL TRIAL: NCT04965480
Title: Detecting Delayed Discharge in Acute Geriatric Unit Using Natural Language Processing
Acronym: COLATERAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0153
Record Dates: First submitted 2021-07-08; First posted 2021-07-16 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Language; Geriatric; Older; Electronic Health Record
Keywords: Natural Language Process; appropriate stay; acute geriatric unit; older; Electronic Health Record.
MeSH Terms: conditions — Language

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delayed discharge in geriatric units is a health and economic issue. There is no algorithm to automatically measure the appropriateness of admissions or hospital days. 30% of the days of hospitalization in acute geriatric units (AGU) are not appropriate. Waiting for a transfer to a follow-up care and rehabilitation unit (SSR) is the main risk factor for inappropriate days. The purpose of this project is to develop an algorithm using natural language processing to predict the appropriateness of an admission to UGA, or a day at UGA.

ELIGIBILITY:
Inclusion Criteria:

* age : >75 years
* patient hospitalized in an AGU

Exclusion Criteria:

* refusal to participate

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged >75 years, hospitalized in AGU in Amiens University Hopsital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Concordance between Appropriateness Evaluation Protocol algorithm prediction result and real admission in AGU | 15 days
  AGU is acute geriatric units
Concordance between Appropriateness Evaluation Protocol algorithm prediction result and real admission for one day in AGU | one day
  AGU is acute geriatric units

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No